CLINICAL TRIAL: NCT06684483
Title: Quantifying Associations of Stress and Inflammation-Associated Oral Biomarkers With Oral Health, Oral Health Behaviors, Systemic Biomarkers and Clinical Phenotype in Individuals With Alcohol Use Disorder (AUD)
Brief Title: The Impact of Heavy Alcohol Use on Saliva and Oral Health
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10002005; 002005-CC
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12-04

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence
Keywords: Oral Health Behaviors; Alcohol Use Disorder; Salivary Bioscience; Stress; Health Behaviors; Salivary Biomarker; Inflammation; Neuropsychological Symptoms
MeSH Terms: conditions — Alcoholism; Health Behavior; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Age, smoking status and gender matched healthy volunteers.
- Patients with AUD: Patients with alcohol use disorder seeking inpatient treatment.

SUMMARY:
Background:

People with alcohol use disorder (AUD) have a higher rate of dental and gum disease. Poor oral health can increase the risk of other diseases, such as diabetes and stroke. Researchers want to learn more about how to identify developing inflammation in the mouth. They also want to know how improved oral health education and behaviors can affect inflammation in people with AUD.

Objective:

This study has 2 goals: (1) to test the usefulness of a new questionnaire about oral health and (2) to learn more about how oral health behaviors affect inflammation in people with AUD.

Eligibility:

People aged 18 years and older who are staying on an inpatient unit being treated for AUD. Healthy volunteers are also needed.

Design:

The study is divided into 2 parts: People will participate in either one part or the other.

In part 1, participants will have 1 visit. They will have a physical exam. They will answer 18 questions for a survey about how they care for their teeth.

In part 2, participants with AUD will have a physical exam. They will provide saliva and blood samples. They will have a dental exam with X-rays. They will fill out questionnaires about their health, mental health, social habits, diet, and sleep. They will keep a diary of their nicotine use for 4 weeks while inpatient.

Healthy volunteers will have 1 visit. They will have a physical exam and provide blood and saliva samples. They will have a dental exam with X-rays. They will fill out questionnaires.

DETAILED DESCRIPTION:
Study Description:

This is an observational pilot protocol aimed at exploring relationships between clinical phenotype, subjective oral health behaviors, objective oral health, salivary/oral biomarkers, and blood biomarkers in treatment-seeking individuals with alcohol use disorder (AUD). This study has two parts: Part 1 will consist of cognitive interviews to evaluate the content validity and interpretability of the Oral Health Behaviors Assessment Questionnaire (OHBA). Part 2 will include collecting biological and behavioral data including saliva samples, oral mouthwash samples, blood samples, dental exams, and health behavior and symptom data using instruments including the OHBA. The aims of Part 2 are to evaluate the feasibility of salivary biospecimen collection in the quantification of oral and systemic stress and inflammation-associated biomarkers in patients with AUD, and to produce preliminary data for associations of specific oral biomarkers with objective oral health, oral health behaviors, systemic biomarkers, and clinical phenotype in patients with AUD compared to controls matched on age, sex, and smoking status.

Objectives:

Part 1

Primary Objective:

To evaluate the interpretability and construct validity of the OHBA by conducting cognitive interviews in both treatment-seeking participants with AUD and healthy control participants.

Part 2

Primary Objectives:

* To evaluate study procedures in using saliva samples to measure inflammation and stress-associated biomarkers in participants with AUD and controls.
* To examine relationships between oral health behaviors, oral health, clinical symptoms, salivary characteristics, salivary biomarkers, and blood biomarkers in patients with AUD and controls.

Secondary Objectives:

* To assess the impact of heavy alcohol consumption on salivary characteristics and salivary biomarkers in treatment-seeking patients with AUD at inpatient admission versus controls.
* To evaluate if oral health, salivary characteristics, and salivary biomarkers change as patients undergo inpatient treatment for AUD.

To determine if associations between oral health, salivary characteristics, salivary biomarker levels, blood biomarker levels, and clinical symptoms differ after a period of abstinence from alcohol as patients undergo inpatient treatment for AUD (i.e., within-group comparison of admission visit versus dental exam visit).

Tertiary/Exploratory Objectives:

* To explore correlations and measure differences between oral microbiome-associated biomarkers and oral health, salivary characteristics, salivary biomarker levels, blood biomarker levels, and clinical symptoms in patients with AUD and controls.
* To determine if associations between oral microbiome characteristics and oral health, salivary characteristics, salivary biomarker levels, blood biomarker levels, and clinical symptoms differ after a period of abstinence from alcohol as patients undergo inpatient treatment for AUD.

Endpoints:

Part 1

Primary Endpoint:

Completion of cognitive interviewing, research team meeting to discuss results and editing of any language in the OHBA (if applicable) based on the cognitive interviewing results used to improve subject understanding and acceptability of the questions in the instrument. Submission of OHBA revisions to IRB will be made if edits to the instrument are made.

Part 2

Primary Endpoints:

* Feasibility (sample processing, saliva characterization, analyte measurement and analysis considerations) of saliva biomarker quantification measured after two visits in patients with AUD (admission visit, dental exam visit) and one visit in controls (dental exam visit).
* Quantification of oral health behaviors, oral health, clinical symptoms, salivary characteristics (salivary flow rate, salivary pH) and salivary and blood biomarker levels in patients with AUD and controls at dental exam visit.

Secondary Endpoints:

* Quantification of oral health (Modified Beck's Oral Assessment Scale [Modified BOAS], dental exam assessment metrics), clinical symptoms (perceived stress, anxiety, depression, and sleep disturbance), salivary characteristics (salivary flow rate, salivary pH) in patients with AUD at inpatient admission visit and controls at dental exam visit.
* Changes in oral health, salivary characteristics, and salivary biomarker levels in patients with AUD from admission visit to dental exam visit.
* Changes in relationships between oral health, salivary characteristics, and salivary biomarker levels with blood biomarker levels, and clinical symptoms in patients with AUD from admission visit to dental exam visit.

Tertiary/Exploratory Endpoints:

* Quantification of oral microbiome community characteristics in patients with AUD and controls at dental exam visit. Measurement of relationships between oral microbiome characteristics with oral health behaviors, oral health, clinical symptoms, salivary characteristics, and salivary and blood biomarker levels in patients with AUD and controls at dental exam visit.
* Differences in oral microbiome community characteristics in patients with AUD from admission visit to dental exam visit. Changes in relationships between oral microbiome community characteristics with oral health, salivary characteristics, and salivary biomarker levels with blood biomarker levels, and clinical symptoms in patients with AUD from admission visit to dental exam visit.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

AUD participants:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Treatment-seeking individuals aged 18 years or older.
* Able to read and speak English.
* Admitted and consented for 14-AA-0181 at the NIH CC for inpatient treatment.
* Part 1 Only: Agree for audio recording of cognitive interview.
* Part 2 Only: BMI less than or equal to 30 kg/m^2.

Healthy Control Participants:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Individuals aged 18 years or older.
* Able to read and speak English.
* Self-reported to be in good physical health.
* Part 1 Only: Agree for audio recording of cognitive interview.
* Part 2 Only: BMI less than or equal to 30 kg/m^2.
* AUDIT score of 7 or below.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

Patients with AUD and Healthy Control Participants:

* The presence of a condition or illness that would hamper the individual giving informed consent (e.g., cognitive impairment).
* Part 2 Only: Self-reported presence of a condition or illness that would prevent the individual to have a diagnostic oral examination (e.g., oral cancer of the mouth, Sjogren's syndrome).
* Part 2 Only: Currently taking or have taken any of the following medications within the last month by self-report; Antibiotics, Corticosteroids, Immunosuppressive or Cytotoxic agents. Topical antibiotics and/or corticosteroids on areas other than the oral cavity are not exclusion criteria.
* Pregnant or breastfeeding
* Subjects who participate in Part 1 of the protocol will not be eligible for Part 2.
* Non-English speakers: we do not have a Spanish version of OHBA, and we are exploring cognitive interviewing of the instrument in English currently. Also, the pt's on 1SE (half of the focused population for this study) are not typically Spanish speakers. We also do not have many of the surveys we plan to administer in Spanish, and they may not be available in other languages.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part 1 of the study will recruit adults (>=18 years) who are enrolled in inpatient treatment for AUD (n=6) and healthy controls (n=6) to conduct cognitive interviews and evaluate the interpretation of the Oral Health Behaviors Assessment measure. Part 2 will recruit adults (>=18 years) who are enrolled in inpatient treatment for AUD at the NIH Clinical Center (n=30) and healthy controls matched on age, sex, and smoking status (n=30). The total sample size of this study, including both Parts 1 and 2 participants will be n=72.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of a total of 12 cognitive interviews in participants with AUD (n=6) & healthy participants (n=6). Editing of any language in the OHBA (if applicable) as a result of the cognitive interviewing results. | Until endpoint is reached.
  The endpoint will refine the OHBA questionnaire, if needed, to improve subject understanding and acceptability of the questions in the instrument; a primary measure in the Part 2 portion of the current study.
Feasibility of saliva biomarker quantification measured after 2 visits in patients with AUD and one dental visit in controls. | When recruitment and sample processing is complete.
  This endpoint will identify if salivary samples are appropriate to measure inflammation and stress-associated biomarkers in patients with AUD, if special procedures need to be performed to quantify salivary biomarkers in patients with AUD and the identification of other variables that may influence salivary samples in patients with AUD for future research consideration.
Quantification of oral health behaviors, oral health, clinical symptoms, salivary characteristics, and salivary and blood biomarker levels in patients with AUD and controls at dental exam visit. | When recruitment and sample processing is complete.
  The endpoints will be measured to evaluate relationships between potential salivary signaling biomarkers and multiple facets of oral and systemic health and health behaviors.

SECONDARY OUTCOMES:
Quantification of oral health, clinical symptoms, salivary characteristics in patients with AUD at inpatient admission visit and controls at dental exam visit. | When recruitment and sample processing is complete.
  Comparison of saliva characteristics and associated biomarkers shortly after a period of heavy alcohol use in patients with AUD compared to controls.
Changes in oral health, salivary characteristics, and salivary biomarker levels in patients with AUD from admission visit to dental exam visit | When recruitment and sample processing is complete.
  This will allow evaluation if saliva characteristics and associated biomarkers change during a period of abstinence from alcohol after heavy use in patients with AUD.
Changes in relationships between oral health, salivary characteristics, and salivary biomarker levels with blood biomarker levels, and clinical symptoms in patients with AUD from admission visit to dental exam visit. | When recruitment and sample processing is complete.
  Assessment if there is a difference in associations between oral health and salivary characteristics with blood biomarker levels and clinical symptoms when evaluated in the context of heavy alcohol use compared to a period of sobriety in the same population during inpatient treatment for AUD.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Maki, C.R.N.P., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be deposited into a data repository in line with NIH regulations.
Supporting Information: SAP, Analytic Code
Time Frame: In line with publication of results.
Access Criteria: De-identified datasets used to generate results presented in manuscripts will be deposited into a repository that can be publicly accessible in line with NIH regulations. In compliance with ethical standards and institutional policies, other access to individual participant data will be governed by a structured data-sharing framework to ensure participant privacy and confidentiality. Access to IPD will be granted under a Data Use Agreement that specifies permissible uses, prohibits re-identification or further data sharing, and requires secure storage and handling of data. Access will be restricted to de-identified or coded datasets, with direct identifiers removed.

REFERENCES:
- [Background] Maki KA, Ganesan SM, Meeks B, Farmer N, Kazmi N, Barb JJ, Joseph PV, Wallen GR. The role of the oral microbiome in smoking-related cardiovascular risk: a review of the literature exploring mechanisms and pathways. J Transl Med. 2022 Dec 12;20(1):584. doi: 10.1186/s12967-022-03785-x. PMID 36503487
- [Background] Barb JJ, Maki KA, Kazmi N, Meeks BK, Krumlauf M, Tuason RT, Brooks AT, Ames NJ, Goldman D, Wallen GR. The oral microbiome in alcohol use disorder: a longitudinal analysis during inpatient treatment. J Oral Microbiol. 2021 Dec 1;14(1):2004790. doi: 10.1080/20002297.2021.2004790. eCollection 2022. PMID 34880965
- [Background] Maki KA, Crayton CB, Butera G, Wallen GR. Examining the relationship between the oral microbiome, alcohol intake and alcohol-comorbid neuropsychological disorders: protocol for a scoping review. BMJ Open. 2024 Mar 21;14(3):e079823. doi: 10.1136/bmjopen-2023-079823. PMID 38514150
- [Derived] Maki KA, Xu S, Wallen GR, Gerrard C, Sung C, Papneja S, Tuason RTS, Ramchandani VA, Diazgranados N, Barb JJ. Associations between oral health behaviours, oral health, salivary biomarkers and clinical phenotype in individuals with alcohol use disorder: protocol for a longitudinal observational study. BMJ Open. 2025 Dec 17;15(12):e101197. doi: 10.1136/bmjopen-2025-101197. PMID 41407429
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002005-CC.html